CLINICAL TRIAL: NCT04544033
Title: IL- 6 Gene (174G/C) Single Nucleotide Polymorphism as an Indicator of COVID-19 Severity in Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, bsant safwat kasem, principle investigator, Tanta University
Other Study IDs: IL6 in egyptian COVID patients
Record Dates: First submitted 2020-09-05; First posted 2020-09-10 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample will be collected on EDTA containing tubes. Peripheral blood sample will be collected on plain tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild group: Amendment to MOH COVID-19 Protocol:
  * Patient with mild clinical symptoms & clinically table.
  * CT changes: Appearance in the lung from no changes to just subpleural nodule or subpleural line.
  Interventions: Diagnostic Test: interleuken 6 level measurment; Diagnostic Test: Interleukin-6 Gene-174C detection
- moderate group: Amendment to MOH COVID-19 Protocol:
  * Patient with non-specific and specific respiratory infection (pneumonia).
  * CT changes in both lungs (Ground glass opacities (GGO), Crazy paving, consolidation, multiple interlobular thickening).
  Interventions: Diagnostic Test: interleuken 6 level measurment; Diagnostic Test: Interleukin-6 Gene-174C detection
- severe group: Amendment to MOH COVID-19 Protocol:
  * Patients with respiratory distress (RR > 30/min, Sa02 < 92 at room air).
  * Chest radiology showing more than 50% lesion or progressive lesion within 24 to 48 hours.
  * CT changes in both lungs: extensive (GGO, Crazy paving, consolidation, multiple interlobular thickening, fan shaped distribution of peribronchial thickening).
  Interventions: Diagnostic Test: interleuken 6 level measurment; Diagnostic Test: Interleukin-6 Gene-174C detection

INTERVENTIONS:
Diagnostic Test: interleuken 6 level measurment — Detection of IL6 level using ELISA technique.
Diagnostic Test: Interleukin-6 Gene-174C detection — The genotyping of the polymorphisms in IL-6 promoter G-174C (rs1800795) will be performed using PCR-RFLP technique.

SUMMARY:
Although the direct damage from the viruses contributes to the initiation of the disease, the cytokine storm caused by COVID-19 plays a vital role in the development of acute lung injury and adult respiratory distress syndrome. IL-6, a kind of pleiotropic cytokine, is expressed by immune cells such as DC, monocytes, macrophages, B cells, and subsets of activated T cells, as well as by non-immune cells like fibroblasts, epithelial cells, and keratinocytes

DETAILED DESCRIPTION:
The World Health Organization (WHO) declared coronavirus disease 2019 (COVID-19) a public health emergency of international concern the epidemic has put public health systems under severe strain both in western countries and in the developing world. SARS-CoV-2 displays a more efficient transmission pattern when compared with SARS-CoV and MERS-CoV. Although the direct damage from the viruses contributes to the initiation of the disease, the cytokine storm caused by COVID-19 plays a vital role in the development of acute lung injury and adult respiratory distress syndrome.

IL-6, a kind of pleiotropic cytokine, is expressed by immune cells such as DC, monocytes, macrophages, B cells, and subsets of activated T cells, as well as by non-immune cells like fibroblasts, epithelial cells, and keratinocytes. It contributes to the pathogenesis of inflammatory or autoimmunity diseases. Excessive production of IL-6 leads to serious disease progression in viral infection. The IL-6 gene is located on chromosome 7 and several polymorphisms have been reported. The most frequently studied polymorphism is the single nucleotide polymorphism (SNP) 174C and - 174G in the promoter region, which has been associated with transcription rates of IL6. The incidence of IL-6-174C alleles is approximately 40%among the general Population. The G allele 174 SNP is coupled with the increased transcription upon endotoxin and IL-1β stimulation, IL-6 -174C allele carrier status is associated with higher level of IL-6 production and more severe forms of 4 pneumonia in general. This analysis strengthens the notion that IL-6 plays a pivotal role in novel coronavirus pneumonia (NCP) progression, it was IL-6-174 C allele rather than G allele that contributed to the risk of sepsis induced by Pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Patients proved to be COVID-19 positive
* clinical correlation with positive PCR.
* clinical correlation with positive rapid antigen detection test.

Exclusion Criteria:

* Patients with chronic infections including hepatitis B or C infection.
* Immunodeficiency virus (HIV) infections.
* Autoimmune diseases including systemic lupus erthromatosus and rheumatoid arthritis.
* Any malignancy or chronic inflammation
* Any other chest diseases (TB)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients proved to be COVID-19 positive by clinical correlation with positive PCR or rapid antigen detection test.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
interleuken- 6 gene (174G/C) single nucleotide polymorphism | "through study completion, an average of 4 months
  the correlation between IL- 6 gene (174G/C) single nucleotide polymorphism with the pathogenesis of COVID-19 severity in Egyptian patients.

SECONDARY OUTCOMES:
interleukin 6 level | "through study completion, an average of 4 months
  the correlation between IL-6 with the pathogenesis of COVID-19 severity in Egyptian patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Bsant Safwat Kasem, Tanta, El Gharbyia, Egypt